CLINICAL TRIAL: NCT02030769
Title: Pronase Improves Efficacy of Chromoendoscopy Screening on Esophageal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Collaborators: Beijing Tide Pharmaceutical Co., Ltd (Industry)
Responsible Party: Principal Investigator, Zhiguo Liu, Associate Professor, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20130925-4
Record Dates: First submitted 2014-01-06; First posted 2014-01-09 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Esophageal Neoplasms
Keywords: Esophageal Neoplasms; Lugol's solution; Pronase; Endoscopy, Digestive System; Pretreatment method
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Pronase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pronase (Experimental): Add pronase 20000 U in 80ml pretreatment mixture plus 5ml Dimethicone and 1g sodium bicarbonate.
  Interventions: Drug: Pronase
- control (Sham Comparator): No pronase in 80ml pretreatment mixture plus 5ml Dimethicone and 1g sodium bicarbonate.
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Pronase — use pronase to improve visibility during endoscopical iodine staining
  Arms: Pronase
Drug: Control — No pronase plus Dimethicone and sodium bicarbonate. use without pronase to compare visibility during endoscopical iodiine staining
  Arms: control

SUMMARY:
Lugol's solution staining was regarded as a gold standard to detect early superficial lesion during esophageal cancer screening using endoscopy. However, the sensitivity and specificity were influenced by mucus and food debris of esophagus. Pronase, a kind of protease, was previously shown to improve the visibility of gastrointestinal tract. It's unknown if the pre-treatment with pronase would also improve the quality of iodine staining in esophagus.A randomized double-blind clinical trial was designed to investigate whether or not pronase might improve detection rate of early esophageal lesion, especially high grade dysplasia and early cancer by improving the esophageal visibility.

ELIGIBILITY:
Inclusion Criteria:

* Patients 60 years to 75 years old
* Patients less than 60 years old, but with one or multiple high risk factors for esophageal cancer including smoking and drinking addiction,family history of esophageal cancer, personal history of esophageal or head and neck malignancies, previous endoscopy documenting iodine void superficial lesion.

Exclusion Criteria:

* Allergy to iodine or any other medicine which used in this trial.
* Previous endoscopy revealing advanced esophageal cancer or other non-superficial lesions.
* Conditions interfering visibility of endoscope including gastrointestinal obstruction and upper gastrointestinal bleeding.
* Anatomic variation by surgery.
* Pregnancy
* Other conditions which investigator consider the patient at high risk for complications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Detection rate of high grade dysplasia and carcinoma in iodine void lesion | 1 week
  Detection Rate=（lesions with confirmed high grade dysplasia/all iodine void lesions）*100%

SECONDARY OUTCOMES:
Average Esophageal Visibility Score Before iodine staining | 30 min after ingesting pretreatment solution
Average Esophageal Visibility Score After iodine staining | within 5 min after iodine staining
Detection Rate of lesions with pink sign | within 5 min after iodine staining
overall detection rate of iodine void lesion | within 5 min after iodine staining

OTHER OUTCOMES:
observation time for esophagus | with 30 min after intubation

CONTACTS AND LOCATIONS:
Overall Officials: Kaichun Wu, Ph.D. & M.D., Study Chair — Xijing Hospital of Digestive DIsease
Locations (1):
- Xijing Hospital of Digestive Disease, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Lopes AB, Fagundes RB. Esophageal squamous cell carcinoma - precursor lesions and early diagnosis. World J Gastrointest Endosc. 2012 Jan 16;4(1):9-16. doi: 10.4253/wjge.v4.i1.9. PMID 22267978
- [Background] Yokoyama A, Hirota T, Omori T, Yokoyama T, Kawakubo H, Matsui T, Mizukami T, Mori S, Sugiura H, Maruyama K. Development of squamous neoplasia in esophageal iodine-unstained lesions and the alcohol and aldehyde dehydrogenase genotypes of Japanese alcoholic men. Int J Cancer. 2012 Jun 15;130(12):2949-60. doi: 10.1002/ijc.26296. Epub 2011 Sep 16. PMID 21796615
- [Background] Dubuc J, Legoux J-, Winnock M, Seyrig J-, Barbier J-, Barrioz T, Laugier R, Boulay G, Grasset D, Sautereau D, Grigoresco D, Butel J, Scoazec J-, Ponchon T; Societe Francaise d'Endoscopie Digestive. Endoscopic screening for esophageal squamous-cell carcinoma in high-risk patients: a prospective study conducted in 62 French endoscopy centers. Endoscopy. 2006 Jul;38(7):690-5. doi: 10.1055/s-2006-925255. PMID 16874909
- [Background] Ishihara R, Yamada T, Iishi H, Kato M, Yamamoto S, Yamamoto S, Masuda E, Tatsumi K, Takeuchi Y, Higashino K, Uedo N, Tatsuta M, Ishiguro S. Quantitative analysis of the color change after iodine staining for diagnosing esophageal high-grade intraepithelial neoplasia and invasive cancer. Gastrointest Endosc. 2009 Feb;69(2):213-8. doi: 10.1016/j.gie.2008.04.052. Epub 2008 Aug 20. PMID 18718584
- [Background] Shimizu Y, Omori T, Yokoyama A, Yoshida T, Hirota J, Ono Y, Yamamoto J, Kato M, Asaka M. Endoscopic diagnosis of early squamous neoplasia of the esophagus with iodine staining: high-grade intra-epithelial neoplasia turns pink within a few minutes. J Gastroenterol Hepatol. 2008 Apr;23(4):546-50. doi: 10.1111/j.1440-1746.2007.04990.x. Epub 2007 Jun 15. PMID 17573830
- [Derived] Zhao X, Guo M, Zhu S, Zhang L, Dong T, Luo H, Yu W, Zhu J, Fan X, Han Y, Liu Z. Pre-procedure oral administration of pronase improves efficacy of lugol chromoendoscopy in esophageal squamous cell carcinoma screening: a prospective, double-blinded, randomized, controlled trial. Surg Endosc. 2023 Jun;37(6):4421-4430. doi: 10.1007/s00464-023-09902-1. Epub 2023 Feb 13. PMID 36781469